CLINICAL TRIAL: NCT04381286
Title: Transpulmonary Driving Pressure in ARDS COVID19 Patients / TRANSPULMONARY-COVID19
Brief Title: Transpulmonary Driving Pressure in ARDS COVID19 Patients
Acronym: TRANSPULMONARY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0194
Record Dates: First submitted 2020-04-23; First posted 2020-05-08 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Mechanical Ventilation; SARS-CoV-2; COVID-19
Keywords: elastance; Acute respiratory distress syndrome; Esophageal pressure; Pleural pressure
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A majority (65-85%) of critically ill patients admitted in intensive care units with a confirmed diagnostic of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) developed an acute respiratory distress syndrome (ARDS) according to BERLIN criteria. Gattinoni et al. recently described that the ARDS related to SARS-CoV-2 was not a "Typical" ARDS. Patients affected by this infection present indeed a major hypoxemia, which was surprisingly associated in early phase with a high compliance of respiratory system, more than 50 ml/cm H2O in most cases. The cornerstone of current treatment in case of ARDS is the use of "lung protective" ventilation, including limited tidal volumes (VT), low end-inspiratory plateau pressures while maintaining sufficiently-high positive end-expiratory pressures (PEEP). However, high levels of PEEP in patients may have detrimental effects on hemodynamic status and fluid retention, particularly when the respiratory system compliance is normal. High PEEP may also lead to overdistension and an increase of alveolar dead space. The airway pressures commonly monitored does not reliably reflect the impact of pressures on the lung parenchyma. Elastance of chest wall may indeed largely influence values of airways pressions. In contrast, transpulmonary pressure obtained using esophageal pressure (Pes) directly reflect lung overdistension risk and lung properties. In order to better understand this new kind of ARDS characterized by modest recruitable profile and to better personalize mechanical ventilation setting and therapy it is obvious to precise transpulmonary pressure.

ELIGIBILITY:
Inclusion criteria:

* Major patients (18-90 years old)
* Hospitalized following SARS-CoV-2
* Mechanical ventilatory support

Exclusion criteria:

* Minor patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with SARS-CoV-2 and mechanical ventilation requirement
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical Ventilation | 1 day
  Duration of mechanical Ventilation

SECONDARY OUTCOMES:
Number of Participants with during of Acute respiratory distress syndrom (SDRA) | 1 day
  Number of Participants with during of Acute respiratory distress syndrom (SDRA)
Length of stay in intensive care unit | 1 day
  Length of stay in intensive care unit
Mortality | 1 day
  Mortality
number of patients with pulmonary complications | 1 day
  number of patients with pulmonary complications
Number of Participants with pulmonary stress and strain | 1 day
  Number of Participants with pulmonary stress and strain

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Séverin, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC